CLINICAL TRIAL: NCT01009177
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate the Effect of Bosentan in Patients With Stage IV Metastatic Melanoma Treated With Dacarbazine
Brief Title: Effect of Bosentan in Patients With Metastatic Melanoma Treated With Dacarbazine (DTIC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC-052-281
Record Dates: First submitted 2009-10-14; First posted 2009-11-06 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Melanoma
Keywords: Melanoma; Metastatic; DTIC; Bosentan
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bosentan (Experimental)
  Interventions: Drug: Bosentan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosentan — Bosentan 500 mg bid
  Arms: Bosentan
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study is designed as a multicenter, double blind, parallel-group, placebo-controlled, randomized, event driven Phase II study of DTIC with or without bosentan as first-line treatment in patients with stage IV melanoma.

DETAILED DESCRIPTION:
This is a randomized, double-blind (1:1 bosentan : placebo) trial to evaluate the effect of bosentan in combination with DTIC on TTP or death in patients with metastatic melanoma stage IV.

The patients will receive study medication (bosentan or placebo) and DTIC for 35 weeks to 105 weeks; the study will be completed when 66 events (tumor progression, death due to underlying disease, other/additional anti-tumor therapy) have been observed.

Study drug will be administered orally, 500 mg twice a day. DTIC will be given once every three weeks in a dosage of 1000 mg/m2 intravenously (i.v.) or in accordance with the Institution's DTIC treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years of age or older
2. Histologically proven malignant melanoma (Balch et al., J. Clin Oncol. 19(16): 3635-48, 2001) with stage IV measurable disease as defined by RECIST criteria (Therasse et al., J Natl Cancer Inst, 92(3): 205-16, 2000).
3. Patients with prior radiation therapy (> 30 days prior to study drug initiation) will be allowed provided the indicator lesion(s) used for this study was (were) outside the field of radiation or represent new lesions not previously irradiated.
4. Patients who had no prior therapy with DTIC.
5. Patients with cutaneous melanoma lesions must consent to having a biopsy obtained during the screening period and at the end of treatment for exploratory analysis of endothelin receptor expression. Biopsies obtained prior to the study that have been frozen in accordance with procedures specified for this protocol may be used.
6. ECOG performance status (≤ 2)
7. Life expectancy > 12 weeks
8. Female patients must be non-pregnant, non-breast feeding, and either post menopausal, surgically sterile, or practicing a reliable method of contraception (hormonal methods alone are not sufficient)
9. Provide written informed consent
10. Willing to return to study center for follow up

Exclusion Criteria:

1. ALT and/or AST > 3 × the upper limit of normal (ULN) at screening OR ALT and /or AST > 2 x ULN and total bilirubin > 2.0 mg/dl at screening
2. Lactate dehydrogenase > 1.5 x ULN
3. Hemoglobin >30% below the lower limit of normal
4. Systolic blood pressure < 85 mmHg
5. NYHA class III/IV congestive heart failure
6. Any prior chemotherapy, biological therapy or immunotherapy for stage IV metastatic disease.
7. Received immunotherapy < 30 days before treatment start (completed adjuvant immunotherapy for previous resected metastatic disease is allowed)
8. Concurrent use of calcineurin inhibitors (cyclosporine A, tacrolimus), sirolimus, fluconazole or glibenclamide (glyburide) or expected to receive any of these drugs during the study at inclusion and during the study.
9. History of other malignancy in the last 5 years, with the exception of squamous cell carcinoma of the skin treated with local resection and basal cell carcinoma
10. CNS metastases or carcinomatous meningitis
11. Ocular melanoma
12. Known hypersensitivity to any excipients of Tracleer™
13. Prior therapy with bosentan
14. Use of therapy with another investigational drug within 4 weeks of the start of dosing with bosentan or plan to receive such treatment during the study
15. Known drug or alcohol dependence or any other factor that will interfere with the conduct of the study
16. Any standard contraindications for the use of DTIC as per Australian package insert

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Time to tumor progression (TTP) or death (progression free survival) after initiation of treatment. Tumor progression is defined per RECIST criteria. | 6 weekly

SECONDARY OUTCOMES:
• Tumor response rate • Duration of overall response • Best overall response • Survival will be assessed at 12 months after initiation of study drug and every year thereafter for 5 years | 6 weekly

CONTACTS AND LOCATIONS:
Overall Officials: Andjela Kusic-Pajic, MD, Study Director — Actelion Pharmaceuticals Australia Pty. Ltd

REFERENCES:
- [Derived] Kefford RF, Clingan PR, Brady B, Ballmer A, Morganti A, Hersey P. A randomized, double-blind, placebo-controlled study of high-dose bosentan in patients with stage IV metastatic melanoma receiving first-line dacarbazine chemotherapy. Mol Cancer. 2010 Mar 30;9:69. doi: 10.1186/1476-4598-9-69. PMID 20350333